CLINICAL TRIAL: NCT01904409
Title: A Randomized, Double-blind, Placebo-controlled, Dose-ranging, Multicenter Study to Assess the Efficacy and Safety of Rifaximin Soluble Solid Dispersion (SSD) Tablets for the Prevention of Complications in Subjects With Early Decompensated Liver Cirrhosis
Brief Title: Dose-ranging Study of Rifaximin Soluble Solid Dispersion (SSD) Tablets for the Prevention of Complications of Early Decompensated Liver Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RNLC2131
Record Dates: First submitted 2013-07-17; First posted 2013-07-22 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Rifaximin; Serine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo (Placebo Comparator): Placebo tablets once daily.
  Interventions: Drug: Placebo
- Rifaximin SSD 40 mg IR tablet (Experimental): Rifaximin soluble solid dispersion (SSD) 40 mg immediate release (IR) tablet once daily.
  Interventions: Drug: Rifaximin SSD 40 mg IR tablet
- Rifaximin SSD 80 mg IR tablet (Experimental): Rifaximin soluble solid dispersion (SSD) 80 mg immediate release (IR) tablet once daily.
  Interventions: Drug: Rifaximin SSD 80 mg IR tablet
- Rifaximin SSD 40 mg SER tablet (Experimental): Rifaximin soluble solid dispersion (SSD) 40 mg sustained extended release (SER) tablet once daily.
  Interventions: Drug: Rifaximin SSD 40 mg SER tablet
- Rifaximin SSD 80 mg SER tablet (Experimental): Rifaximin soluble solid dispersion (SSD) 80 mg sustained extended release(SER) tablet once daily.
  Interventions: Drug: Rifaximin SSD 80 mg SER tablet
- Rifaximin SSD 80mgIR/80mgSER tablet (Experimental): Rifaximin soluble solid dispersion (SSD) 80 mg immediate release (IR) tablet + rifaximin SSD 80 mg sustained extended release (SER) tablet once daily.
  Interventions: Drug: Rifaximin SSD 80mgIR/80mgSER tablet

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: Rifaximin SSD 40 mg IR tablet
  Other Names: Rifaximin
  Arms: Rifaximin SSD 40 mg IR tablet
Drug: Rifaximin SSD 80 mg IR tablet
  Other Names: Rifaximin
  Arms: Rifaximin SSD 80 mg IR tablet
Drug: Rifaximin SSD 40 mg SER tablet
  Other Names: Rifaximin
  Arms: Rifaximin SSD 40 mg SER tablet
Drug: Rifaximin SSD 80 mg SER tablet
  Other Names: Rifaximin
  Arms: Rifaximin SSD 80 mg SER tablet
Drug: Rifaximin SSD 80mgIR/80mgSER tablet
  Other Names: Rifaximin
  Arms: Rifaximin SSD 80mgIR/80mgSER tablet

SUMMARY:
The primary objective of this study is to assess the efficacy of rifaximin SSD versus placebo in preventing complications of liver cirrhosis, such as all-cause mortality (death due to all causes) or hospitalization, in subjects with early decompensated liver cirrhosis.

Rifaximin, a non-systemic antibacterial agent, is currently marketed as a 550 mg tablet for the reduction in risk of recurrent overt hepatic encephalopathy, a complication of liver cirrhosis. The rifaximin SSD tablet was formulated to maximize the efficacy of rifaximin.

Subjects will receive 1 of 5 doses of rifaximin SSD tablets or placebo tablets every day for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of liver cirrhosis and documented ascites.
* Model End Stage Liver Disease (MELD) score of at least 12, MELD Na of at least 12, or Child-Pugh B (score of 7 - 9).
* If applicable, has a close family or other personal contacts who can provide continuing oversight to the patient and will be available to the patient during the conduct of the trial.
* If female of childbearing potential, have a negative serum pregnancy test at study start and agree to use an acceptable method of contraception during the study.

Exclusion Criteria:

* History of a major psychiatric disorder including uncontrolled major depression or controlled or uncontrolled psychoses within the past 24 months prior to study start.
* History of alcohol abuse or substance abuse within the past 3 months prior to study start.
* Documented cholestatic liver disease such as primary sclerosing cholangitis.
* Had prophylactic variceal banding within 2 weeks or is scheduled to undergo prophylactic banding during the study.
* Diagnosed with an infection for which the patient is currently taking oral or parenteral antibiotics.
* Significant hypovolemia, or any electrolyte abnormality that can affect mental function (eg, serum sodium < 125 mEq/L, serum calcium > 10 mg/dL).
* Severe hypokalemia, defined as serum potassium concentration < 2.5 mEq/L.
* Anemic, defined as hemoglobin concentration ≤ 8 g/dL.
* Renal insufficiency with a creatinine of ≥ 1.5 mg/dL.
* Presence of intestinal obstruction or inflammatory bowel disease.
* Uncontrolled Type 1 or Type 2 diabetes.
* History of seizure disorders.
* Unstable cardiovascular or pulmonary disease, categorized by a worsening in the disease condition that requires a change in treatment or medical care within 30 days of study start.
* Active malignancy within the last 5 years (exceptions: basal cell carcinomas of the skin, or if female, in situ cervical carcinoma that has been surgically excised).
* Has hepatocellular carcinoma.
* Known human immunodeficiency virus, varicella, herpes zoster, or other severe viral infection within 6 weeks of study start.
* Positive stool test for Yersinia enterocolitica, Campylobacter jejuni, Salmonella, Shigella, ovum and parasites, and/or Clostridium difficile (C. difficile); determined during the screening period prior to study start.
* History of tuberculosis infection and/or has received treatment for a tuberculosis infection.
* History of hypersensitivity to rifaximin, rifampin, rifamycin antimicrobial agents, or any of the components of rifaximin soluble solid dispersion.
* Used any investigational product or device, or participated in another research study within 30 days prior to study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Time to all-cause mortality or hospitalization that is attributable to complications of liver disease. | Weeks 1 through 24
  The primary outcome measure will evaluate the time from start of the treatment period to death due to any cause (all-cause mortality) or hospitalization due to complications of liver disease for each patient during the 24-week treatment period.

SECONDARY OUTCOMES:
Overall hospitalization rate due to each complication of liver disease or all-cause mortality over the 24-week treatment period. | Weeks 1 through 24
  This outcome measure will determine the rate of hospitalization (percentage of patients who are hospitalized) due to each complication of liver disease or all-cause mortality over the 24-week treatment period.
Pharmacokinetics of rifaximin and its metabolite. | Weeks 1 through 24
  This outcome will measure the plasma levels of rifaximin and its metabolite (25-desacetyl rifaximin) for each patient during the 24-week treatment period.
Incidence of treatment-emergent adverse events. | Weeks 1 through 24
  This outcome will evaluate the incidence of treatment-emergent adverse events (percentage of patients who experience adverse events following the start of the treatment period).
Change in clinical laboratory parameters. | Weeks 1 through 24
  This outcome will measure the changes in each patient's clinical laboratory test results during the treatment period.
Changes in electrocardiogram measurements | Weeks 1 through 24
  This outcome will measure the changes in measurements obtained from 12-lead electrocardiograms for each patient during the treatment period.
Changes in indices of health outcomes | Weeks, 4, 8, 12, 16, and 24
  This outcome will evaluate each patient's responses on questionnaires that assess health status.

CONTACTS AND LOCATIONS:
Overall Officials: James Joffrion, Study Director — Bausch Health Americas, Inc.
Locations (110):
- United States (103):
  - Salix Investigative Site, Birmingham, Alabama
  - Salix Investigative Site, Dothan, Alabama
  - Salix Investigative Site, Mobile, Alabama
  - Salix Investigative Site, Tucson, Arizona
  - Salix Investigational Site, Artesia, California
  - Salix Investigational Site, Bakersfield, California
  - Salix Investigational Site, Chula Vista, California
  - Salix Investigational Site, Coronado, California
  - Salix Investigational Site, Costa Mesa, California
  - Salix Investigative Site, Fresno, California
  - Salix Investigational Site, La Jolla, California
  - Salix Investigative Site, Los Angeles, California
  - Salix Investigational Site, Monterey, California
  - Salix Investigational Site, Riverside, California
  - Salix Investigational Site, San Diego, California
  - Salix Investigational Site, Ventura, California
  - Salix Investigational Site, Englewood, Colorado
  - Salix Investigational Site, Littleton, Colorado
  - Salix Investigational Site, Bristol, Connecticut
  - Salix Investigational Site, New Haven, Connecticut
  - Salix Investigational Site, Waterbury, Connecticut
  - Salix Investigational Site, Coral Gables, Florida
  - Salix Investigational Site, Gainesville, Florida
  - Salix Investigative Site, Hialeah, Florida
  - Salix Investigational Site, Hialeah, Florida
  - Salix Investigational Site, Hollywood, Florida
  - Salix Investigative Site, Inverness, Florida
  - Salix Investigational Site, Lake Worth, Florida
  - Salix Investigative Site, Largo, Florida
  - Salix Investigative Site, Maitland, Florida
  - Salix Investigational Site, Miami, Florida
  - Salix Investigational Site, Miami Springs, Florida
  - Salix Investigational Site, New Port Richey, Florida
  - Salix Investigative Site, Orlando, Florida
  - Salix Investigational Site, Pembroke Pines, Florida
  - Salix Investigational Site, Port Orange, Florida
  - Salix Investigational Site, Saint Cloud, Florida
  - Salix Investigational Site, Tamarac, Florida
  - Salix Investigational Site, Atlanta, Georgia
  - Salix Investigative Site, Atlanta, Georgia
  - Salix Investigative Site, Decatur, Georgia
  - Salix Investigational Site, Macon, Georgia
  - Salix Investigative Site, Chicago, Illinois
  - Salix Investigative Site, Maywood, Illinois
  - Salix Investigational Site, Evansville, Indiana
  - Salix Investigational Site, Indianapolis, Indiana
  - Salix Investigative Site, Iowa City, Iowa
  - Salix Investigational Site, Bowling Green, Kentucky
  - Salix Investigational Site, Bastrop, Louisiana
  - Salix Investigational Site, Monroe, Louisiana
  - Salix Investigational Site, New Orleans, Louisiana
  - Salix Investigational Site, Shreveport, Louisiana
  - Salix Investigational Site, Annapolis, Maryland
  - Salix Investigational Site, Baltimore, Maryland
  - Salix Investigational Site, Chevy Chase, Maryland
  - Salix Investigational Site, Hagerstown, Maryland
  - Salix Investigational Site, Boston, Massachusetts
  - Salix Investigational Site, Brockton, Massachusetts
  - Salix Investigational Site, Springfield, Massachusetts
  - Salix Investigative Site, Chesterfield, Michigan
  - Salix Investigational Site, Wyoming, Michigan
  - Salix Investigational Site, Minneapolis, Minnesota
  - Salix Investigative Site, Tupelo, Mississippi
  - Salix Investigational Site, Kansas City, Missouri
  - Salix Investigative Site, St Louis, Missouri
  - Salix Investigational Site, Marlton, New Jersey
  - Salix Investigational Site, New Brunswick, New Jersey
  - Salix Investigative Site, Brooklyn, New York
  - Salix Investigational Site, Flushing, New York
  - Salix Investigational Site, New York, New York
  - Salix Investigational Site, Rochester, New York
  - Salix Investigative Site, The Bronx, New York
  - Salix Investigational Site, Asheville, North Carolina
  - Salix Investigational Site, Chapel Hill, North Carolina
  - Salix Investigative Site, Charlotte, North Carolina
  - Salix Investigational Site, Charlotte, North Carolina
  - Salix Investigational Site, Fayetteville, North Carolina
  - Salix Investigational Site, Wilmington, North Carolina
  - Salix Investigational Site, Winston-Salem, North Carolina
  - Salix Investigative Site, Cincinnati, Ohio
  - Salix Investigational Site, Cincinnati, Ohio
  - Salix Investigational Site, Cleveland, Ohio
  - Salix Investigative Site, Dayton, Ohio
  - Salix Investigational Site, Mentor, Ohio
  - Salix Investigational Site, Portland, Oregon
  - Salix Investigative Site, Bristol, Tennessee
  - Salix Investigational Site, Chattanooga, Tennessee
  - Salix Investigational Site, Nashville, Tennessee
  - Salix Investigative Site, Arlington, Texas
  - Salix Investigational Site, Austin, Texas
  - Salix Investigational Site, Dallas, Texas
  - Salix Investigative Site, Dallas, Texas
  - Salix Investigational Site, Fort Worth, Texas
  - Salix Investigational Site, Houston, Texas
  - Salix Investigational Site, San Antonio, Texas
  - Salix Investigational Site, Bountiful, Utah
  - Salix Investigative Site, Salt Lake City, Utah
  - Salix Investigational Site, Charlottesville, Virginia
  - Salix Investigative Site, Norfolk, Virginia
  - Salix Investigative Site, Richmond, Virginia
  - Salix Investigational Site, Richmond, Virginia
  - Salix Investigative Site, Richland, Washington
  - Salix Investigative Site, Seattle, Washington
- Russia (7):
  - Salix Investigative Site, Krasnogorsk
  - Salix Investigative Site, Moscow
  - Salix Investigative Site, Novosibirsk
  - Salix Investigative Site, Saint Petersburg
  - Salix Investigative Site, Samara
  - Salix Investigative Site, Smolensk
  - Salix Investigative Site, Stavropol

REFERENCES:
- [Derived] Zacharias HD, Kamel F, Tan J, Kimer N, Gluud LL, Morgan MY. Rifaximin for prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD011585. doi: 10.1002/14651858.CD011585.pub2. PMID 37467180
- [Derived] Bajaj JS, Hassanein TI, Pyrsopoulos NT, Sanyal AJ, Rahimi RS, Heimanson Z, Israel RJ, Rockey DC. Dosing of Rifaximin Soluble Solid Dispersion Tablets in Adults With Cirrhosis: 2 Randomized, Placebo-controlled Trials. Clin Gastroenterol Hepatol. 2023 Mar;21(3):723-731.e9. doi: 10.1016/j.cgh.2022.05.042. Epub 2022 Jun 22. PMID 35750249